CLINICAL TRIAL: NCT05772338
Title: National, Multicenter, Randomized, Double-blind, Pilot Study to Evaluate the Efficacy and Safety of BNP105 in the Treatment of Recurrent Aphthous Stomatitis
Brief Title: Efficacy and Safety of BNP105 in the Treatment of Recurrent Aphthous Stomatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BNP105-P-0123
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-02

CONDITIONS: Aphthous Stomatitis
Keywords: Aphthous Stomatitis
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BNP105 (25 + 25 + 15) (Experimental): Up to six applications per day. The number of drops varies according to the ulcer diameter: 1 to 3 mm: 1 drop; 3 to 6 mm: 2 drops; greater than 6 mm: 3 drops.
  Interventions: Drug: BNP105 (25 + 25 + 15)
- Placebo (Placebo Comparator): Up to six applications per day. The number of drops varies according to the ulcer diameter: 1 to 3 mm: 1 drop; 3 to 6 mm: 2 drops; greater than 6 mm: 3 drops.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BNP105 (25 + 25 + 15) — BNP105 oral suspension, 25 mg + 25 mg + 15 mg, oral. Up to six applications per day.
  Arms: BNP105 (25 + 25 + 15)
Other: Placebo — Placebo. Up to six applications per day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BNP105 in the treatment of recurrent aphthous stomatitis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Age greater than or equal to 12 years;
* One minor recurrent aphthous stomatitis with onset of symptoms within 48 hours;
* Moderate to severe baseline pain, with VAS ≥ 60 mm (EVA scale 0-100 mm).

Exclusion Criteria:

* Any clinical findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participants diagnosed with: Behcet's disease, rheumatoid arthritis, systemic lupus erythematosus, reactive arthritis, Reiter's syndrome, Crohn's disease, ulcerative colitis);
* Participants with diseases that affect healing (e.g. diabetes);
* Immunocompromised participants;
* Participants with aphthous herpetiform ulceration or major aphthous ulceration;
* Participants using medication to treat oral ulcerations (systemic or local);
* Participants who used analgesics or anti-inflammatory drugs in the 6 hours prior to the beginning of the study;
* Participants who used systemic antibiotics in the 2 weeks prior to the beginning of the study;
* Participants using medications that can confuse pain assessment (psychotropics, antidepressants and sedative-hypnotics), except when on a stable dose for at least 30 days prior to the screening visit, and the dose cannot be changed during the clinical trial;
* Participants with current smoking habits.
* Participants who are pregnant, breastfeeding or planning to get pregnant or female participants with the potential to become pregnant who are not using a reliable method of contraception;
* Known hypersensitivity to the formula components used during the clinical trial;
* Participants with current or medical history of cancer in the last 5 years;
* Participants who participated in other research protocol in the last 12 months, unless the investigator judges that there may be a direct benefit to it.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To assess the change in pain intensity after the first application. | 3 and 10 minutes
  Difference in pain intensity 3 and 10 minutes after the first application of the medication compared to baseline, measured by the VAS scale. The VAS consists of a 100 mm line, with two end points representing 0 ("no pain") and 100 (Worst Possible Pain").

SECONDARY OUTCOMES:
To assess the change in pain intensity after 3 days of treatment. | 3 days
  Difference in pain intensity after 3 days of treatment compared to baseline. Pain intensity will be evaluated by the Visual Analogue Scale (VAS). The VAS consists of a 100 mm line, with two end points representing 0 ("no pain") and 100 (Worst Possible Pain").
To assess the pain intensity daily after breakfast, lunch and dinner. | 7 days
  Pain intensity will be evaluated daily after breakfast, lunch and dinner by the Numeric Pain Rating Scale (NPRS). The NPRS is an 11-point scale scored from 0-10 representing 0 ("no pain") and 10 (Worst Possible Pain").
To assess the pain intensity daily at night. | 7 days
  Pain intensity will be evaluated daily at night by the Numeric Pain Rating Scale (NPRS). The NPRS is an 11-point scale scored from 0-10 representing 0 ("no pain") and 10 (Worst Possible Pain").
To assess the oral health-related quality of life | 7 days
  The oral health-related quality of life will be evaluated daily at night by the adapted Oral Health Impact Profile (OHIP) questionary.
Percentage of participants healed after 3 days of treatment. | 3 days
  Percentage of participants healed after 3 days of treatment, defined as ulcer diameter = 0 mm and pain intensity = 0, measured by the VAS scale. The VAS consists of a 100 mm line, with two end points representing 0 ("no pain") and 100 (Worst Possible Pain").
Percentage of participants with no pain after 3 days of treatment. | 3 days
  Percentage of participants with no pain after 3 days of treatment, defined as pain intensity = 0, measured by the VAS scale. The VAS consists of a 100 mm line, with two end points representing 0 ("no pain") and 100 (Worst Possible Pain").
Global assessment of treatment by participant after 3 days of treatment | 3 days
  The global evaluation of the treatment after 3 days of treatment will be evaluated by the categorical scale of 5 points representing 0 = very bad, 1 = bad, 2 = indifferent, 3 = good and 4 = very good.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - EMS, Hortolândia, São Paulo
  - Cecip Jau - Centro de Estudos Clinicos Do Interior Paulista Ltda, Jaú, São Paulo

IPD SHARING:
Plan to Share IPD: No